CLINICAL TRIAL: NCT06150755
Title: Evaluation of Marginal Bone Loss of Two Immediately Loaded Implants Retaining Mandibular Overdentures With Ball Attachment Versus Intra Oral Welding Titanium Bar a Randomized Clinical Trial
Brief Title: Evaluation of Marginal Bone Loss of Two Immediately Loaded Implants Retaining Mandibular Overdenture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Abdelfatah, associate professor of oral and maxillofacial prosthodontics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RecID032118
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Intervention Model Description: completely edentulous patients treated with overdenture retained by immediately loaded implant in the canine region
Who Masked: Outcomes Assessor
Masking Description: Blinding will be done by the outcomes assessor and one of the study authors will remove the prosthetic part before measuring crestal bone loss by outcome assessor through cone paralling technique. Blinding of the outcomes assessor for assessment by oral health questionnaire will be done as well
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mplant supported overdenture by ball attachment (Placebo Comparator): immediate loaded implant supported overdenture by ball attachment
  Interventions: Procedure: implant supported overdenture by ball
- implant supported overdenture by bar (Active Comparator): immediate loaded implant supported overdenture by intraoral welding titanium bar splinted two implant
  Interventions: Procedure: implant supported overdenture by bar

INTERVENTIONS:
Procedure: implant supported overdenture by ball — overdenture supported by two implant with ball attachment
  Arms: mplant supported overdenture by ball attachment
Procedure: implant supported overdenture by bar — overdenture supported by two implant splinted by intraoral welding titanuim bar
  Arms: implant supported overdenture by bar

SUMMARY:
It is a randomized control clinical trial in which maxillary and mandibular dentures will be constructed, two implants will be inserted in the inter foraminal region in the edentulous mandible and immediate loading will be done. We will be comparing peri-implant marginal bone loss of two immediately loaded implants retaining mandibular overdentures with ball attachment versus intra oral welding titanium bar. Patient satisfaction will be assessed using oral health related quality of life.

DETAILED DESCRIPTION:
The patients will be divided in two groups, each group will receive maxillary and mandibular conventional heat cured acrylic resin complete dentures, which will be duplicated and provided by radio-opaque resin at the proposed implant sites to act as radiographic stents. Only patients with a D2 or D3 bone density will be included in the study. This will be confirmed by their cone beam computed tomographic (CBCT) scans of the mandible, while wearing radiographic stents.

The CBCT will be used to ensure sufficient bone width at the proposed implant sites, namely canine regions for implant diameter 3.7. Diagnostic set ups for all patients will be prepared to ensure a crown height space of at least 12 mm to accommodate the ball attachments for group I and intra oral welding bar for group II. Each group will receive two implants in the canine region through using surgical stent and immediate loading will be done.

Group B: immediate loading will be done using ball attachment and soft liners acting as female part for mandibular overdenture.

Group I: immediate loading will be done using intra oral welding titanium bar with 2 mm diameter and soft liner acting as a female part for mandibular overdenture.

For each group, marginal bone loss around the implants will be assessed at time of denture delivery and six months later. Patient satisfaction will be assessed using oral health related quality of life using (OHRQOL 14)

Study population

Patients' selection:

Fifty four edentulous patients will be selected from the out-patient clinic of Removable prosthodontics department, Faculty of Dentistry, Ain Shams University according to inclusion and exclusion criteria. This research will be reviewed by the research ethics committee faculty of dentistry Ain Shams University

Patients' approval:

* All patients will be informed in details about the nature of the investigation and the aim of the study. When they will agree to take part in the study, they will sign on an informed consent form.
* All participants will be given notice about their privacy practices, their legal duties and their rights.
* In case of implant treatment failure, the patients will receive a new well- fitting denture.

Study procedure

Patients' history:

* Medical history: patients will be asked about their medical and dental history through a direct interview and a detailed questionnaire sheet.
* Dental history: patients will be asked about the cause, the date of teeth extraction and if there is any previous experience with any prosthetic appliance, any problems with TMJ will also be recorded.

Patients' examination:

- Extra oral examination:

It will be carried-out to detect any facial abnormalities, signs of inflammation and TMJ disorders as pain, clicking and limited mouth opening as well as maximum opening.

- Intra-oral examination:

Visual examination of the denture bearing area with no flabby tissues, mucous membrane of the cheeks, lips, palate and tongue. They will be checked for no ulceration or signs of inflammation also exclude bony protuberance presence.

Radiographic evaluation and surgical guide construction:

* A panoramic x-ray of the patients preoperatively to determine if the patient is indicated for implant placement.
* Complete denture fabrication for each patient and duplication of the lower one using barium sulphate acrylic resin material to obtain radio opaque stent appliance
* A cone beam computed tomography (CBCT) scan of the patients wearing radiographic stent to evaluate the bone height, width, and density in the canine region.

Randomization and allocation concealment:

Patients will be selected randomly. The method requires the preparation of opaque sealed envelopes, containing the letter "B" and the letter "I" to represent ball attachment and the bar attachment groups respectively.

Patients will be selected according to inclusion and exclusion criteria.

Surgical procedures:

* infiltration anesthesia will be given bilaterally in the canine regions and a crestal incision will be attempted, extending from canine premolar area of one side to that of the other side. This will be done in both groups
* The flap will then be elevated and reflected using a periosteal elevator. The canine areas will be identified by the aid of the surgical guide.
* Drilling will be continued then Implants will be first hand threaded and then threaded using the torque wrench and hex tool 1.25. A minimum insertion torque of 30 Ncm is required to allow for immediate loading.
* Once the implant platform will be flushed with the crestal bone, ball abutment will be attached to the implant for group B and abutment for group I then intraoral welding will be done using 2mm titanium.
* The flap will be sutured using interrupted suturing technique.

Prosthetic insertion

* The mandibular denture will be prepared for the relining procedures by creating sufficient space in the fitting surface of the denture opposite to the attachments.
* Mollosil liner will be used to act as the female receptacle of the ball attachments in group B and intra oral welding titanium bar for group I.
* Patients will be given the following post-insertion instructions; In the first 72 hours it will be recommended to remove the denture only during oral and denture hygiene procedures. Strict oral hygiene measures should be followed by the patient..

ELIGIBILITY:
Inclusion Criteria:

* good oral hygiene
* patient will be medically free
* sufficient inter arch space

Exclusion Criteria:

* heavy smoker
* TMJ disorders
* uncontrolled diabetes
* flappy tissue

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-12-24 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
marginal bone loss measurement | 6 months
  marginal bone loss will be measured mesial and distal to the implant by radiographic cone paralling technique

SECONDARY OUTCOMES:
patient satisfaction | 6 months
  patient satisfaction will be measured by oral health of quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed MA Mohamed, BDS MSc MD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt